CLINICAL TRIAL: NCT01797367
Title: Pulmonary Substudy: A Substudy of Strategic Timing of AntiRetroviral Treatment (START)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0603M83587-4
Record Dates: First submitted 2013-01-22; First posted 2013-02-22 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; HIV
Keywords: HIV; COPD; FEV1; respiratory function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out if starting anti-retroviral therapy (ART) above 500 cluster-of-differentiation-4 (CD4)+ cells/milliliter (mL) ('early ART group') slows the rate of decrease in lung function over time compared to waiting to start ART until the CD4+ drops below 350 cells/mL ('deferred ART group'). Lung function normally declines with age, and both human immunodeficiency virus (HIV) infection and ART have been shown to case a decline in lung function as well. Decline in lung function can be an early indicator of chronic obstructive pulmonary disease (COPD), a significant cause of sickness and death in people with HIV. In this study, lung function will be measured at baseline and every year thereafter by using a spirometer.

ELIGIBILITY:
Inclusion Criteria:

* Simultaneous co-enrollment in the START study
* Signed informed consent to the Pulmonary Substudy
* Age >= 25 years

Exclusion Criteria:

* An episode of respiratory illness with 2 or more symptoms of cough, wheezing, breathlessness, or increase in sputum production within the 6 weeks before baseline spirometry.
* Use of asthma medications (bronchodilator, inhaled corticosteroid, leukotriene inhibitor, or theophylline) for 2 or more consecutive weeks within the 6 months before baseline spirometry.
* Relative contraindications to spirometry, such as chest or abdominal or eye surgery within the 3 months before baseline spirometry, known retinal detachment at the time of baseline spirometry.
* Known allergy to albuterol/salbutamol
* Relative contraindications to albuterol/salbutamol, such as resting heart rate of >110 beats per minute, or a known serious or recurrent or uncontrolled cardiac condition (such as unstable coronary artery disease, decompensated heart failure, or recurrent tachyarrhythmias).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollees are HIV-positive, antiretroviral-naive individuals with CD4+ > 500 cells/mL randomized to the START trial.
Sampling Method: Non-Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2010-03; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in post-bronchodilator forced expiratory volume in 1 second (FEV1) | baseline, then at annual visits for up to 6 years
  FEV1 is measured by having the participant inhale a dose of bronchodilator (albuterol/salbutamol), wait 15 minutes, and then inhale maximally and exhale maximally and forcefully into a spirometer. Participants do at least 3 trials of spirometry for each measurement, and up to 8, to obtain 3 usable measurements.

SECONDARY OUTCOMES:
Change from baseline in respiratory health status using the St. George's Respiratory Questionnaire for COPD (SGRQ-C) | baseline, then at annual visits for up to 6 years
  The SGRQ-C is a standardized, validated, self-administered questionnaire that measures respiratory health status and includes domains of respiratory symptoms, activity limitations, and psychosocial impact. It will be given to participants to complete in their native language. It contains 40 items and takes approximately 10-15 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Ken M Kunisaki, MD, Study Chair — Minneapolis Veterans Affairs Medical Center; Dennis E Niewoehner, MD, Study Chair — University of Minnesota; John E Connett, PhD, Study Chair — University of Minnesota
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] MacDonald DM, Samorodnitsky S, Wendt CH, Baker JV, Collins G, Kruk M, Lock EF, Paredes R, Poongulali S, Weise DO, Winston A, Wood R, Kunisaki KM; INSIGHT START Pulmonary Substudy Group. Pneumoproteins and biomarkers of inflammation and coagulation do not predict rapid lung function decline in people living with HIV. Sci Rep. 2023 Mar 23;13(1):4749. doi: 10.1038/s41598-023-29739-x. PMID 36959289
- [Derived] Hodgson S, Griffin TJ, Reilly C, Harvey S, Witthuhn BA, Sandri BJ, Kunisaki KM, Wendt CH. Plasma sphingolipids in HIV-associated chronic obstructive pulmonary disease. BMJ Open Respir Res. 2017 Apr 3;4(1):e000180. doi: 10.1136/bmjresp-2017-000180. eCollection 2017. PMID 28409005
- [Derived] Kunisaki KM, Niewoehner DE, Collins G, Aagaard B, Atako NB, Bakowska E, Clarke A, Corbelli GM, Ekong E, Emery S, Finley EB, Florence E, Infante RM, Kityo CM, Madero JS, Nixon DE, Tedaldi E, Vestbo J, Wood R, Connett JE; INSIGHT START Pulmonary Substudy Group. Pulmonary effects of immediate versus deferred antiretroviral therapy in HIV-positive individuals: a nested substudy within the multicentre, international, randomised, controlled Strategic Timing of Antiretroviral Treatment (START) trial. Lancet Respir Med. 2016 Dec;4(12):980-989. doi: 10.1016/S2213-2600(16)30319-8. Epub 2016 Oct 20. PMID 27773665
- [Derived] Kunisaki KM, Niewoehner DE, Collins G, Nixon DE, Tedaldi E, Akolo C, Kityo C, Klinker H, La Rosa A, Connett JE; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Pulmonary function in an international sample of HIV-positive, treatment-naive adults with CD4 counts > 500 cells/muL: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 0):119-28. doi: 10.1111/hiv.12240. PMID 25711330
- See also: INSIGHT network website, including information on the START Pulmonary Substudy — http://www.insight-trials.org